CLINICAL TRIAL: NCT04091256
Title: Evaluate Efficacy of Desensitizing Toothpaste Containing Zinc-carbonate Hydroxyapatite Before and After: A 8 Week Clinical Study
Brief Title: Treatment of Tooth Sensitivity With the Use of Biorepair Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Muhammad Khalil Khan, Associate Professor, Qassim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST/55/2019
Record Dates: First submitted 2019-07-26; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Dentinal Hypersensitivity
Keywords: Biorepair sensitive toothpaste; Clinical trial; Dentinal Hypersensitivity; Schiff Sensitivity Scale; Zinc-carbonate hydroxyapatite nanocrystals

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm: Participants will be treated with desensitizing toothpaste containing zinc-carbonate hydroxyapatite nanocrystals (Zn-CHA) for 8 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical trials with a single arm (Experimental): : Participants will be treated with desensitizing toothpaste containing zinc-carbonate hydroxyapatite nanocrystals (Zn-CHA) for 8 weeks.
  Interventions: Other: Single arm clinical study

INTERVENTIONS:
Other: Single arm clinical study — Participants will be treated with desensitizing toothpaste containing zinc-carbonate hydroxyapatite nanocrystals (Zn-CHA) for 8 weeks.

SUMMARY:
The purpose of this clinical study is to evaluate the effect of desensitizing toothpaste containing zinc-carbonate hydroxyapatite nanocrystals in reducing or controlling DH after 8 weeks of treatment

DETAILED DESCRIPTION:
This clinical study design is an 8-week single center, before and after use of desensitize dentifrice. This study will conducted in the College of Dentistry Qassim University. 72 patients surfing from DH, include in the study fulfill the inclusion criteria. All subjects 20 to 70 years of age in good health, and must have 2 teeth with DH, will be included in this study. Screening will be performed for the selection of patients, which fulfill the inclusion criteria. Baseline data will be recorded and Sensitivity was assessed by air-blast sensitivity, using Schiff Sensitivity Scale (SSS).

Sensitivity was assessed by air-blast sensitivity, using Schiff Sensitivity Scale (SSS) described as follows.

0 = Subject does not respond to air stimulus

1. = Subject responds to air stimulus but does not request discontinuation of stimulus
2. = Subject responds to air stimulus and requests discontinuation or moves from stimulus
3. = Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus

ELIGIBILITY:
Inclusion Criteria:

* All male and female subjects 20 to 70 years of age
* All subjects in good health
* All subjects must have 2 teeth with DH, only incisors, canine and premolars were included with the exposed cervical dentin (facial surfaces).

All participants of the study having Schiff Sensitivity Scale score of 2 & 3

Exclusion Criteria:

* Subjects with deep carious teeth, defective restorations
* Any pathological lesion
* Periodontal disease, mobile teeth, cracked enamel, orthodontic appliances,
* Periodontal pockets >4mm
* Subjects using pain control medicines, sensitive toothpaste
* Pregnant or lactating women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Dentine hypersensitivity (DH) evaluation by means of air-blast sensitivity test, using Schiff Sensitivity Scale (SSS) after 4 weeks. | 4 Weeks
  This will be assessed using Schiff Sensitivity Scale (SSS) score difference from the baseline, that will be determined immediately before product use and then after 4 weeks of daily brushing with the test sensitive toothpaste. Tooth sensitivity score was assessed by air-blast sensitivity, using Schiff Sensitivity Scale (SSS) as follows: 0 = Subject does not respond to air stimulus, 1 = Subject responds to air stimulus but does not request discontinuation of stimulus, 2 = Subject responds to air stimulus and requests discontinuation or moves from stimulus, 3 = Subject responds to air stimulus, considers stimulus to be painful, and requests.

SECONDARY OUTCOMES:
Dentine hypersensitivity (DH) evaluation by means of air-blast sensitivity test, using Schiff Sensitivity Scale (SSS) after 8 weeks | 8 Weeks
  This will be assessed using Schiff Sensitivity Scale (SSS) score difference from the baseline, that will be determined immediately before product use and then after 8 weeks of daily brushing with the test sensitive toothpaste. Tooth sensitivity score was assessed by air-blast sensitivity, using Schiff Sensitivity Scale (SSS) as follows: 0 = Subject does not respond to air stimulus, 1 = Subject responds to air stimulus but does not request discontinuation of stimulus, 2 = Subject responds to air stimulus and requests discontinuation or moves from stimulus, 3 = Subject responds to air stimulus, considers stimulus to be painful, and requests.

CONTACTS AND LOCATIONS:
Overall Officials: Dhafer Al Asmari, Board, Principal Investigator — Qassim University; Muhammad K Khan, PhD, Principal Investigator — Qassim University
Locations (1):
- College of Dentistry Qassim University, Buraidah, Al Qassim, Saudi Arabia